CLINICAL TRIAL: NCT06682988
Title: A Randomized Phase 2, Open-label Study of Mirvetuximab Soravtansine in Patients With Platinum-resistant Advanced High-grade Epithelial Ovarian, Primary Peritoneal, or Fallopian Tube Cancers With High Folate Receptor-alpha Expression Testing 2 Schedules of Administration for Dose Optimization, With a Separate Cohort to Determine Starting Dose in Patients With Moderate Hepatic Impairment
Brief Title: A Study to Assess Adverse Events and Change in Disease Activity in Participants With Platinum-Resistant Advanced High-Grade Epithelial Ovarian, Primary Peritoneal, or Fallopian Tube Cancers With High Folate Receptor-Alpha Expression Treated With Intravenously (IV) Infused Mirvetuximab Soravtansine
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMGN853-0425
Record Dates: First submitted 2024-11-08; First posted 2024-11-12 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Advanced High-Grade Epithelial Ovarian; Primary Peritoneal; Fallopian Tube Cancers; High Folate Receptor-Alpha Expression; Platinum Resistant
Keywords: Advanced High-Grade Epithelial Ovarian; Primary Peritoneal; Fallopian Tube Cancers; High Folate Receptor-Alpha Expression; Platinum Resistant; Mirvetuximab Soravtansine; MIRV; IMGN853
MeSH Terms: conditions — Fallopian Tube Neoplasms | interventions — mirvetuximab soravtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Randomized Phase 2 Cohort: Arm A (Experimental): Participants will receive Mirvetuximab Soravtansine at the standard dose on Day 1 of a 21-day cycle.
  Interventions: Drug: Mirvetuximab Soravtansine
- Randomized Phase 2 Cohort: Arm B (Experimental): Participants will receive Mirvetuximab Soravtansine at a lower dose than the standard dose on Day 1 and Day 15 of a 28-day cycle .
  Interventions: Drug: Mirvetuximab Soravtansine
- Hepatic Impairment Cohort : Mirvetuximab Soravtansine (Experimental): Participants will receive Mirvetuximab Soravtansine on Day 1 of a 21-day cycle. Different doses will be given to groups of patients to identify a safe and effective dose.
  Interventions: Drug: Mirvetuximab Soravtansine

INTERVENTIONS:
Drug: Mirvetuximab Soravtansine — intravenous (IV) infusion
  Other Names: MIRV; IMGN853

SUMMARY:
Cancer is a condition where cells in a specific part of body grow and reproduce uncontrollably. The purpose of this study is to assess the safety and efficacy of for Mirvetuximab Soravtansine in participants with platinum-resistant advanced high-grade epithelial ovarian, primary peritoneal, or fallopian tube cancer (platinum-resistant ovarian cancer) (PROC) whose tumors express a high level of folate receptor alpha (FRα).

Mirvetuximab Soravtansine (MIRV) is an investigational antibody drug conjugate designed to selectively kill cancer cells. The antibody (protein) part of MIRV targets tumors by delivering a cell-killing drug to cancer cells carrying a protein called folate receptor alpha (FRα). There are 2 cohorts in this study, the Randomized Phase 2 Cohort and the Hepatic Impairment Cohort. In the Randomized Phase 2 Cohort, participants are placed in 1 of 2 groups, called treatment arms. Each treatment arm receives MIRV on a different schedule (on day 1 every 21 days or on days 1 and 15 every 28 days). The Hepatic Impairment Cohort is designed to determine the starting dose of MIRV in patients with moderately abnormal liver function. Around 110 participants will be enrolled in the study at approximately 75 sites worldwide.

The total study duration will be approximately 24 months.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic and may require frequent medical assessments, blood tests, and scans.

ELIGIBILITY:
Inclusion Criteria:

Both Cohorts

* Participants with a confirmed diagnosis of high-grade serous epithelial ovarian cancer (EOC), primary peritoneal cancer, or fallopian tube cancer.
* Participants with platinum-resistant disease:

  * Participants with 1 prior line of platinum-based therapy who have received ≥ 4 cycles of platinum and had a response (complete response (CR) or partial response (PR)) followed by radiological progressive disease (PD) between > 3 months and ≤ 6 months after the date of the last dose of platinum.
  * Participants with 2 or 3 prior lines of platinum-based therapy who had radiological PD

    * 6 months after the date of the last dose of platinum.
* Participants with progression diagnosed radiographically on or after their most recent line of therapy.
* Participants with an Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1.
* Participants with ≥ 1 lesion that meets the definition of measurable disease by RECIST v1.1 (radiologically measured by the investigator).
* Participants with a tumor that is positive for folate receptor alpha (FRα) expression as determined by the Ventana folate receptor 1 (FOLR1) assay (≥ 75% of tumor staining at 2+ intensity).

Exclusion Criteria:

Both Cohorts

* Participants with endometrioid, clear cell, mucinous, or sarcomatous histology; mixed tumors containing any of the above histologies; or low-grade or borderline ovarian tumor.
* Participants with primary platinum-refractory disease, defined as disease that did not respond (complete response (CR) or partial response (PR)) or that progressed radiographically within 3 months of the last dose of first-line platinum-containing chemotherapy.
* Participants with serious concurrent illness or clinically relevant active infection as outlined in the protocol
* Participants with a history of hemorrhagic or ischemic stroke within 6 months prior to randomization.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-05-28 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Randomized Phase 2 Cohort: Percentage of Participants with Grade >= 2 Treatment-Emergent Corneal Adverse Events (AEs) | Up to Approximately 24 months
  An AE is any noxious, pathologic, or unintended change in anatomical, physiologic, or metabolic function as indicated by physical signs, symptoms, or laboratory changes occurring in any phase of a clinical study, whether or not considered study drug related.
Randomized Phase 2 Cohort: Objective response rate (ORR) | Up to Approximately 24 months
  ORR is defined as best response of confirmed complete response (CR) or partial response (PR), as assessed by the Investigator according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1).
Hepatic Impairment Cohort: Maximal Concentration (Cmax) of Mirvetuximab Soravtansine | Up to Approximately 24 months
  Cmax of MIRV
Hepatic Impairment Cohort: Area Under the Plasma Concentration (AUC) of Mirvetuximab Soravtansine | Up to Approximately 24 months
  AUC of MIRV
Hepatic Impairment Cohort: Trough Concentration (Ctrough) of Mirvetuximab Soravtansine | Up to Approximately 24 months
  Ctrough of MIRV
Hepatic Impairment Cohort: Volume of Distribution at Steady State (Vss) of Mirvetuximab Soravtansine | Up to Approximately 24 months
  Vss) of MIRV
Hepatic Impairment Cohort: Time to Maximal Concentration (Tmax) of Mirvetuximab Soravtansine | Up to Approximately 24 months
  Tmax of MIRV
Hepatic Impairment Cohort: Terminal Half-Life (t1/2) of Mirvetuximab Soravtansine | Up to Approximately 24 months
  t1/2 of MIRV

SECONDARY OUTCOMES:
Randomized Phase 2 Cohort: Percentage of Participants with Treatment-Emergent All-Grade Ocular AEs, Grade >= 2 Peripheral Neuropathy, All-Grade Infusion Reactions, and All-Grade Pneumonitis | Up to Approximately 24 months
  An AE is any noxious, pathologic, or unintended change in anatomical, physiologic, or metabolic function as indicated by physical signs, symptoms, or laboratory changes occurring in any phase of a clinical study, whether or not considered study drug related.
Randomized Phase 2 Cohort: Duration of Response (DOR) as Assessed by the Investigator Using RECIST v1.1 | Up to Approximately 24 months
  Defined as the time from initial investigator-assessed response (complete response (CR) or partial response (PR)) until progressive disease (PD) as assessed by the investigator
Randomized Phase 2 Cohort: Progression-Free Survival (PFS) | Up to Approximately 24 months
  PFS is defined as the time from date of randomization until disease progression or death whichever occurs first.
Randomized Phase 2 Cohort: Overall Survival (OS) | Up to Approximately 24 months
  Overall survival is defined as the time from the date of first dose until the date of death from any cause.
Randomized Phase 2 Cohort: Percentage of Participants With CA-125 Confirmed Clinical Response Per Gynecologic Cancer Intergroup (GCIG) Criteria | Up to Approximately 24 months
  The GCIG CA-125 response is defined as at least 50% reduction in CA-125 levels from baseline. The response must be confirmed and maintained for at least 28 days.
Randomized Phase 2 Cohort: Maximal Concentration (Cmax) of Mirvetuximab Soravtansine | Up to Approximately 24 months
  Cmax of MIRV
Randomized Phase 2 Cohort: Area Under the Plasma Concentration (AUC) of Mirvetuximab Soravtansine | Up to Approximately 24 months
  (AUC) of MIRV
Randomized Phase 2 Cohort: Trough Concentration (Ctrough) of Mirvetuximab Soravtansine | Up to Approximately 24 months
  Ctrough of MIRV
Randomized Phase 2 Cohort: Volume of Distribution at Steady State (Vss) of Mirvetuximab Soravtansine | Up to Approximately 24 months
  Vss of MIRV
Randomized Phase 2 Cohort: Time to Maximal Observed Concentration (Tmax) of Mirvetuximab Soravtansine | Up to Approximately 24 months
  Tmax of MIRV
Randomized Phase 2 Cohort: Terminal Half-Life (t1/2) of Mirvetuximab Soravtansine | Up to Approximately 24 months
  t1/2 of MIRV
Randomized Phase 2 Cohort: Change from baseline in two dosing methods while assessing drug response | Up to Approximately 24 months
  Determine the differences in dose amount and exposure between two dosing methods and the effects on exposure-response (ER) relationships
Both Cohorts: Number of Participants With Treatment-emergent Adverse Events (TEAEs) | Up to Approximately 24 months
  An AE is any noxious, pathologic, or unintended change in anatomical, physiologic, or metabolic function as indicated by physical signs, symptoms, or laboratory changes occurring in any phase of a clinical study, whether or not considered study drug related.
Both Cohorts: Percentage of Participants with Clinically Significant Vital Sign Measurements as Assessed by the Investigator | Up to Approximately 24 months
  Vital signs include blood pressure, heart rate, respiratory rate, and body temperature.
Both Cohorts: Percentage of Participants with Clinically Significant Laboratory Values (test) as Assessed by the Investigator | Up to Approximately 24 months
  Percentage of participants with clinically significant laboratory values (hematology, chemistry, and coagulation) as assessed by the investigator.
Both Cohorts: Number of Participants With Clinically Significant Abnormalities in Physical Examination Findings | Up to Approximately 24 months
  Physical examination included assessments of general appearance, skin, head (eyes, ears, nose, and throat), neck, lungs, heart, abdomen, back, lymph nodes, extremities, and neurological system.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (37):
- United States (6):
  - First Physicians Group /ID# 272180, Sarasota, Florida
  - St. Elizabeth Medical Center - Edgewood /ID# 272113, Edgewood, Kentucky
  - Baptist Health Lexington /ID# 272211, Lexington, Kentucky
  - UMass Memorial Medical Center /ID# 272122, Worcester, Massachusetts
  - Karmanos Cancer Institute - Detroit /ID# 272112, Detroit, Michigan
  - Allegheny Health Network West Penn Hospital /ID# 272267, Pittsburgh, Pennsylvania
- Australia (7):
  - Blacktown Hospital /ID# 272182, Blacktown, New South Wales
  - Newcastle Private Hosptial /ID# 272213, Lambton Heights, New South Wales
  - Royal Brisbane and Women's Hospital /ID# 272123, Brisbane, Queensland
  - Icon Cancer Centre Chermside /ID# 272220, Chermside, Queensland
  - Ballarat Base Hospital /ID# 272240, Ballarat, Victoria
  - Monash Health - Monash Medical Centre /ID# 272234, Clayton, Victoria
  - Sir Charles Gairdner Hospital /ID# 272116, Nedlands, Western Australia
- Belgium (3):
  - Algemeen Ziekenhuis klina /ID# 272127, Brasschaat, Antwerpen
  - AZ Maria Middelares /ID# 272186, Ghent, Oost-Vlaanderen
  - AZ-Delta /ID# 272250, Roeselare, West-Vlaanderen
- South Korea (9):
  - National Cancer Center /ID# 272265, Goyang-si, Gyeonggido
  - CHA Bundang Medical Center /ID# 271590, Seongnam, Gyeonggido
  - Seoul National University Bundang Hospital /ID# 271594, Seongnam-si, Gyeonggido
  - Keimyung University Dongsan Hospital /ID# 271592, Daegu, Gyeongsangbuk-do
  - Seoul National University Hospital /ID# 272264, Seoul, Seoul Teugbyeolsi
  - Yonsei University Health System Severance Hospital /ID# 271593, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center /ID# 272130, Seoul, Seoul Teugbyeolsi
  - Gangnam Severance Hospital /ID# 272217, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 271591, Seoul, Seoul Teugbyeolsi
- Spain (9):
  - Hospital Universitario Germans Trias i Pujol /ID# 272216, Badalona, Barcelona
  - Hospital Universitario de Jaén /ID# 272205, Jaén, Jaen
  - Clinica Universidad de Navarra - Pamplona /ID# 275742, Pamplona, Navarre
  - Hospital Universitario Virgen del Rocio /ID# 272107, Seville, Sevilla
  - Hospital Universitario Vall de Hebron /ID# 272134, Barcelona
  - Hospital General Universitario Gregorio Maranon /ID# 272121, Madrid
  - CLINICA UNIVERSIDAD DE NAVARRA-Madrid /ID# 272221, Madrid
  - Hospital Universitario HM Sanchinarro /ID# 272190, Madrid
  - Hospital Clinico Universitario Lozano Blesa /ID# 272165, Zaragoza
- United Kingdom (3):
  - Addenbrookes Hospital /ID# 272162, Cambridge, Cambridgeshire
  - Royal Devon & Exeter Hospital /ID# 272170, Exeter, Devon
  - University College London Hospital /ID# 272115, London, Greater London

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing, visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=IMGN853-0425